CLINICAL TRIAL: NCT00441155
Title: An Extension to a Phase I Multicenter, Dose Escalation Study of Nilotinib in Combination With Imatinib on a Continuous Daily Dosing Schedule in Adult Patients With Imatinib-Resistant Gastrointestinal Stromal Tumors (GIST)
Brief Title: Patients Completing Core Protocol (CAMN107A2103), Exhibiting Stable Disease (SD), Partial Response (PR) or Complete Response (CR) to Nilotinib in Combination With Imatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2103E1
Record Dates: First submitted 2007-02-26; First posted 2007-02-28 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Oncology; Cancer; Imatinib-Resistant Gastrointestinal Stromal Tumors; GIST; Nilotinib; Imatinib-Resistant Gastrointestinal Stromal Tumors (GIST)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasms | interventions — nilotinib; Imatinib Mesylate

ARMS (2):
- Monotherapy: AMN107 (Experimental): initial dose of imatinib (dose level 1) was 400 mg bid was administered orally on a continuous daily schedule and was not escalated during the study
  Interventions: Drug: Nilotinib, Imatinib
- Combination Therapy: AMN107 + Imatinib (Active Comparator): six possible doses of Nilotinib (100 mg once daily (qd), 200 mg qd, 400 mg qd, 200 mg bid, 300 mg bid, and 400 mg bid). four possible doses of Imatinib (0 mg, 400 mg qd, 600 mg qd, and 400 mg bid).the initial dose of nilotinib (dose level 1) was 200 mg qd and could have been escalated up to 400 mg bid
  Interventions: Drug: Nilotinib, Imatinib

INTERVENTIONS:
Drug: Nilotinib, Imatinib — Nilotinib 50 mg and 200 mg gelatin capsules and Imatinib 100 mg and 400 mg film-coated tablets in bottles.. Medication labels for each study drug complied with the legal requirements of each country, were printed in the local language.

SUMMARY:
To provide study drug to patients that benefit from treatment judged by the investigator - to obtain additional long-term safety and efficacy data of this combination regimen in GIST

ELIGIBILITY:
Inclusion criteria:

* Documented Complete Response, Partial Response, or Stable Disease at the time of entry to extension study and/or possible benefit from continuing treatment in the view of the investigator.
* Normal organ and marrow function as defined in core protocol (CAMN107A2103).
* Extension protocol written informed consent.

Exclusion criteria:

* Inability to swallow the medication.
* Any unresolved adverse events related to participation in the core protocol (CAMN107A2103).
* A history of noncompliance to medical regimens or inability or unwillingness to return for all scheduled visits.

Other protocol defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of nilotinib either as single agent or in combination with Imatinib | AE monitored continuously from day 1 cycle 1 to the study completion visit; safety laboratory and cardiac safety monitored every 3 treatment cycles (every 3 months) from day 1 cycle 1 to the study completion visit
  Assessed by AE evaluation, including safety laboratory and cardiac safety (ECG, cardiac enzymes, ECHO) measures.

SECONDARY OUTCOMES:
To assess any clinical responses in Imatinib-resistant GIST patients. Assessment of tumor response will be made based on modified RECIST criteria - to be assessed at the end of every cycle of treatment | every 3 months, at completion of every third treatment cycle prior to first dose of next cycle, at study completion visit
  Assessment of tumor response will be made based on modified RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; NovartisPharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Novartis Investigative Site, Lyon, France
- Novartis Investigative Site, Milan, MI, Italy